CLINICAL TRIAL: NCT05456672
Title: Investigation of the Impact of Food Combination Strategies on Postprandial Blood Glucose Responses
Brief Title: Glycemic Response to Different Food Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Santo Espírito (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Daniela Freitas, Dr, Hospital de Santo Espírito
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GlucoMatchMaker
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Postprandial Glycemia
Keywords: Digestion; Starch; Glycemic Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention (Experimental): Dietary intervention using standardized test meals
  Interventions: Other: Test meals and food baskets

INTERVENTIONS:
Other: Test meals and food baskets — Interventional dietary study using standardized test meals and personalized food baskets to investigate the impact of food combination on the glycemic response. The study period is organized as follows:
  (Day 1: Continuous blood glucose monitoring system (CGM) activation) Days 2 and 3: Two standardized daily menus (breakfast, lunch, afternoon snack and dinner) provided on a randomized crossover basis.
  Days 4 to 7: four standardized test meals, participants will be asked to substitute one meal each day (lunch or dinner) for a test meal according to a pre-defined randomization plan.
  Days 8 to 10: Participants will be asked to prepare all meals using a food basket containing a mix of standardized and personal preference items.
  Days 11 to 13: Participants will be asked to prepare all meals using a food basket containing a mix of standardized and personal preference items and following dietary recommendations developed by the study staff.
  (Day 14: CGM sensor removed)

SUMMARY:
The purpose of this study is to assess the impact of combining starch rich foods with low pH foods on the glycemic response to meals

DETAILED DESCRIPTION:
Low pH foods can attenuate the glycemic response to starch-rich foods. It has been demonstrated that lemon juice, due to its low pH (pH≈2.3) inhibited key digestive enzymes thereby interrupting gastric digestion of starch in vitro. This effect can significantly reduce the glycemic response in humans. In particular, adding lemon juice to a starch rich meal reduced the mean blood glucose concentration peak by 30%.

Considering the panoply of food options available, it is likely that other combinations have similar effects but no work has been conducted to develop a consolidated knowledge base to exploit this strategy. GlucoMatchMaker will go beyond the state-of-the art by addressing this knowledge gap. The main goal is to develop and test the real-life impact of pH-based food combination strategies on glycemic responses.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent
* Subject is available to participate in the study sessions on the proposed dates.

Exclusion Criteria:

* Subject has an allergy or intolerance to any food and/or ingredient in the study meals
* Body mass index ≤ 18.5 kg/m2 or ≥ 30.0 kg/m2.
* Diagnosed mouth, throat or active gastrointestinal pathology that may affect normal ingestion and digestion of food.
* History of pancreatic disease
* Subject is immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year).
* Subject has Type 1 or Type 2 diabetes mellitus or pre-diabetes.
* Subject has a history of drug and/or alcohol abuse at the time of enrolment.
* Subject is currently taking medication that can effect glucose metabolism and/or normal gastrointestinal function.
* Subject is currently participating in another study, or plans to participate in another study during the study period.
* Women of child-bearing potential who do not use an acceptable method of contraception.
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Glycemic response | 12 days
  Measurement of postprandial glucose concentrations

SECONDARY OUTCOMES:
Composition of non standardized meals | 10 days
  Participants' food diaries
Adherence to food combination recommendations | 3 days
  Based on participants' food diaries while using the food baskets provided on days 11 to 13
Salivary alpha-amylase activity | Baseline
  Amylolytic activity of salivary alpha-amylase
AMY 1 copy number | Baseline
  Salivary amylase gene (AMY1) copy number
Dietary patterns | Baseline
  Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Hospital de Santo Espírito da Ilha Terceira, Angra do Heroísmo, Azores
  - TERInov, Angra do Heroísmo, Azores

IPD SHARING:
Plan to Share IPD: No